CLINICAL TRIAL: NCT04235127
Title: The Catalonia Suicide Risk Code Epidemiology Study: a Two-Stage Exposure-Enriched Nested Case-Control Study of Suicide Attempts in Catalonia, Spain
Brief Title: The Catalonia Suicide Risk Code Epidemiology Study: an Epidemiological Study of Suicide Attempts in Catalonia, Spain
Acronym: CSRC-Epi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital del Mar Research Institute (IMIM) (Other)
Collaborators: Catalan Agency for Health Information, Assessment and Quality (Other Government); National Centre for Suicide Research and Prevention, Norway (Unknown); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Jordi Alonso, M.D., Ph.D., Coordinator of the Health Services Research Group, Director of the Epidemiology and Public Health Program, Hospital del Mar Research Institute (IMIM)
Other Study IDs: CSRC-EPI (2017/7431/I)
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Suicide, Attempted; Suicide; Suicide and Self-harm
Keywords: nested case-control study; electronic healthcare records; register-based study; incidence; risk factors; risk prediction; machine learning techniques; inverse probability weighting; public health; surveillance; population-attributable risk proportions
MeSH Terms: conditions — Suicide, Attempted; Suicide; Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Catalan population: The target population consists of the dynamic cohort of all Catalan residents during the 6-year period 2014-2019. Annual total population of Catalonia is between 7.5-7.6 million, with annual rates for immigration, emigration, birth and death being ~2.5%, ~1.9%, ~0.9%, and ~0.8%, respectively. Based on these figures, we expect a maximum of ~9.1 million individuals with Catalan residency status on at least one point in time over the 2014-2019 period. However, we expect SA in Catalonia to be extremely rare before the age of 10, in line with findings that self-injurious behaviour generally occurs as from the adolescent period. We will therefore exclude cases and controls that have not reached age 10 by the end of the 2014-2019 period (i.e., ~10.9%), lowering the total expected target population to ~8.1 million.
  Interventions: Other: sociodemographic variables, somatic conditions, mental disorders, treatment and drug use

INTERVENTIONS:
Other: sociodemographic variables, somatic conditions, mental disorders, treatment and drug use — * sociodemographic variables
  * history of self-injurious behaviours; all types of somatic conditions; neurodevelopmental, mental, behavioural, personality and substance use disorders; all types of medical procedures performed; and number and type of healthcare contacts.
  * prescriptions for psychopharmacological products
  * the Suicidal Scale of the Mini-International Neuropsychiatric Interview, the type and lethality of the attempt that warranted evaluation, presence and type of mental disorder, hopelessness, impulsivity, aggressiveness, altered state of conscience, use or dependence of alcohol, use or dependence of illicit drugs, serious somatic disease (including chronic diseases, chronic pain, and disabilities), living status, presence of family or social support, social problems, stressful life events, access to lethal means, and family history of suicide

SUMMARY:
Suicide attempts (SA) constitute a major public health issue worldwide. Research suggests that 2.7% of adult people ever attempt suicide; among children and adolescents this is estimated to be 6.0%. SA are related to subsequent suicide which represents an annual loss of 34.6 million years of life worldwide. Suicide attempts are also related to persistent physical and mental health issues, psychiatric hospitalizations, impaired academic performance, unemployment, partner abuse victimization and perpetration, having children removed by social services, loneliness, relationship difficulties, impaired social functioning and low life satisfaction. Despite this considerable societal impact, there is a lack of epidemiological research focussing on providing suicide attempt surveillance in the population, to inform public health action aimed at reducing risk for suicide attempts in the population, and to provide data-driven support for suicide risk assessment across healthcare settings. To address this shortcoming, the investigators designed the Catalonia Suicide Risk Code Epidemiology study. Using centralized Electronic Healthcare Record data from the entire public healthcare system of Catalonia, Spain, the CSRC-Epi study aims to estimate reliable suicide incidence rates, identify suicide attempt risk factors, and develop validated suicide attempt risk prediction tools.

ELIGIBILITY:
Inclusion Criteria:

* Catalan residency during 2014-2019
* age 10 or more at end of observation period

Exclusion Criteria:

* none

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population consists of the dynamic cohort of all Catalan residents during the 6-year period 2014-2019.
Sampling Method: Probability Sample
Enrollment: 186000 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of catalan residents with suicide attempt (incidence) | 2014-2019
  Suicide attempt is a nonfatal, self-directed, potentially injurious behaviour with a non-zero degree of intent to die as a result of the behaviour, even if the behaviour does not result in injury

SECONDARY OUTCOMES:
Number of Catalan residents committing suicide (incidence) | 2014-2019
  Suicide is a fatal, self-directed, injurious behaviour with a non-zero degree of intent to die as a result of the behaviour

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mortier P, Vilagut G, Puertolas Gracia B, De Ines Trujillo A, Alayo Bueno I, Ballester Coma L, Blasco Cubedo MJ, Cardoner N, Colls C, Elices M, Garcia-Altes A, Gene Badia M, Gomez Sanchez J, Martin Sanchez M, Morros R, Prat Pubill B, Qin P, Mehlum L, Kessler RC, Palao D, Perez Sola V, Alonso J; CODIRISC Epidemiology Study Group. Catalonia Suicide Risk Code Epidemiology (CSRC-Epi) study: protocol for a population-representative nested case-control study of suicide attempts in Catalonia, Spain. BMJ Open. 2020 Jul 12;10(7):e037365. doi: 10.1136/bmjopen-2020-037365. PMID 32660952
- See also: Related Info — http://www.codirisc.org